CLINICAL TRIAL: NCT06890260
Title: A Clinical Randomized Controlled Study of Electroacupuncture Combined With Microneedle Knife in the Treatment of Moderate to Severe Allergic Rhinitis
Brief Title: The Treatment of Moderate to Severe Allergic Rhinitis With Electroacupuncture Combined With Microneedle Knife
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pengfei Qiu (Other)
Responsible Party: Sponsor-Investigator, Pengfei Qiu, Attending Chinese Medicine Practitioner, Zhejiang Hospital
Organization: Zhejiang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025ZR001
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Allergic Rhinitis (Disorder); Electroacupuncture; Microneedle Knife
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cetirizine hydrochloride tablets combined with nasal budesonide spray group (Experimental): The control group will be given oral cetirizine hydrochloride tablets and nasal budesonide spray with the following dosage: the starting dose is 2 sprays in each nostril twice daily, which is reduced to 1 spray in each nostril twice daily after 3 days, and then change to 1 spray once daily after 1 week, which will be used as the maintenance dose for a total of 4 weeks of treatment.
  Interventions: Drug: Cetirizine hydrochloride tablets combined with nasal budesonide spray.
- Electroacupuncture combined with Microneedle knife group (Experimental): Subjects in this group will be treated with Electroacupuncture combined with Microneedle knife.The treatment time is 30 minutes each time, once every other day, and the treatment is carried out 3 times a week for 4 consecutive weeks, for a total of 12 treatments.
  Interventions: Other: Electroacupuncture combined with Microneedle Knife

INTERVENTIONS:
Other: Electroacupuncture combined with Microneedle Knife — The patient takes the supine position, the acupoints take bilateral Yingxiang acupoints and upper Yingxiang acupoints, the tip of the needle is stabbed obliquely towards the root of the nose for 5-10mm, to the extent that there is a feeling of soreness and distension in the nose, and perform the flat tonic and flat cathartic method, the waveform of electroacupuncture is selected as sparse and dense wave, the frequency is 2/100Hz, the strength of the current is taken as the degree that the patient can tolerate it, and the time of energizing is 30min; and then the patient takes the seated position, with his head hanging down low on the therapeutic pillow, and the therapeutic point of occipitocervical segment is selected, Then the patient is placed on the therapeutic pillow in a sitting position with the head hanging low, the treatment point of the occipitocervical segment is selected, the treatment point of the cervicothoracic junction is marked, and the micro-needle knife cuts and loose
  Arms: Electroacupuncture combined with Microneedle knife group
Drug: Cetirizine hydrochloride tablets combined with nasal budesonide spray. — Cetirizine hydrochloride tablets (specification: 10mg*24 tablets, Suzhou Sinochem Pharmaceutical Industry Co., Ltd., State Pharmaceutical License: H20030447) shall be given, 1 tablet daily. At the same time, nasal budesonide spray (specification: 64μg*120 sprays, AstraZeneca Pharmaceuticals Co., Ltd, State Pharmaceutical License: J20090079) shall be used: the starting dose shall be 2 sprays in each nostril twice a day, and after 3 days, it shall be reduced to 1 spray in each nostril twice a day, and then changed to 1 spray once a day after 1 week, which shall be used as the maintenance dose. The dosage will be increased or decreased at the patient's discretion according to the symptomatic condition during the course of treatment for a total of 4 weeks of treatment and observation. No other drugs for allergic rhinitis will be used during the treatment period.
  Arms: Cetirizine hydrochloride tablets combined with nasal budesonide spray group

SUMMARY:
Based on the inclusion and exclusion criteria, patients with allergic rhinitis who meet the requirements are selected as trial subjects, and the efficacy is clarified in a randomized controlled design trial. We will Use the total nasal symptom score as the primary outcome index, serum chemokine, intercellular adhesion molecule-1, eosinophil cationic protein, total non-nasal symptom score, and rhinitis-related quality of life scale as secondary outcome indexes, and oral cetirizine hydrochloride tablets and nasal budesonide spray as the control group, the efficacy of the subjects in the electroacupuncture combined with microneedle knife group and the drug group will be observed respectively before treatment, after 2 weeks of treatment, after 4 weeks, 1 month follow-up after the end of treatment, and 3 months follow-up after the end of treatment. 4 weeks later, 1 month follow-up after the end of treatment and 3 months follow-up after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Those with clinical and laboratory diagnosis of moderate to severe allergic rhinitis;
2. Aged ≥18 years and ≤75 years, with no restriction on gender or ethnicity;
3. Not taking drugs such as antihistamines or nasal steroids within 1 month before enrollment;
4. Those who voluntarily participated in this study and signed an informed consent form, and who were able to adhere to outpatient treatment for 4 weeks.

Exclusion Criteria:

1. Atrophic rhinitis, hypertrophic rhinitis, vasomotor rhinitis, acute and chronic sinusitis, nasal polyps, severe septal deviation, eosinophilia non-allergic rhinitis;
2. Those with other allergic diseases such as asthma, urticaria, and colds that cause nasal congestion, runny nose, and sneezing;
3. Those who have serious diseases such as cardiovascular, cerebrovascular, hepatic, renal and hematopoietic systems in combination;
4. Pregnant or lactating women, psychiatric patients, patients with malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-11 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score | TNSS will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 3 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale will be performed by two trained raters to perform a Total Nasal Symptom Score#TNSS#, usually in the form of conversation and observation. After the examination, the two raters will score independently.TNSS score of 0 to 16 values, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Total Non-nasal Symptom Score | TNNSS will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 3 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale will be performed by two trained raters to perform a Total Non-nasal Symptom Score#TNNSS#, usually in the form of conversation and observation. After the examination, the two raters will score independently.TNNSS score of 0 to 5 values, and higher scores mean a worse outcome.
Rhinitis Quality of Life Questionnaire | RQLQ will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 3 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale will be performed by two trained raters to perform a Rhinitis Quality of Life Questionnaire Score#RQLQ#, usually in the form of conversation and observation. After the examination, the two raters will score independently.RQLQ score of 0 to 144 values, and higher scores mean a worse outcome.
blood serum | In the early morning at fasting state before and after 4 weeks of treatment
  In both groups, 5 mL of elbow venous blood will be drawn at room temperature in the early morning at fasting state before and after 4 weeks of treatment, and the serum will be separated by centrifugation at 3000 r/min for 15 min, and then stored in a refrigerator at -70℃ for measurement. Serum Eotaxin, Inter Cellular Adhesion Molecule-1(ICAM-1) and Eosinophil Cationic Protein(ECP) expression levels will be measured by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No